CLINICAL TRIAL: NCT00944216
Title: Efficacy and Safety of Salkera Emollient Foam in the Treatment of Moderate to Severe Keratosis Pilaris, a Prospective Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: terminated due to administrative reasons.
Sponsor: Wright State University (Other)
Collaborators: PreCision Dermatology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KP
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Results first posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Keratosis Pilaris
Keywords: keratosis pilaris
MeSH Terms: conditions — Burnett Schwartz Berberian syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Salkera Emollient Foam Treatment (Experimental): All participants will receive this intervention.
  Interventions: Drug: Salkera Emollient Foam

INTERVENTIONS:
Drug: Salkera Emollient Foam — application of the Salkera emollient foam twice a day during the 12 week study period.

SUMMARY:
Keratosis pilaris (KP) is a benign skin condition that often is very frustrating for the patients and treating physicians. The investigators are interested to see if the study product is effective in treating moderate to severe KP.

DETAILED DESCRIPTION:
Keratosis pilaris (KP) is a benign, inherited skin disorder that presents as grouped, rough, horny follicular papules. It is estimated that 40-50% of the adult population and 50-80% of adolescents suffer from KP. Both men and women are affected, with a possible female predominance. It is noted worldwide and shows no racial predilection. Most patients with KP are actually unaware that the condition has a designed medical term. Although no clear etiology had been identified, KP is sometimes associated with other skin conditions such as icththyosis vulgaris, xerosis or atopic dermatitis.

Many patients with KP never seek medical attention since they are asymptomatic. However, KP can create significant cosmetic concerns in some cases. It can also become symptomatic especially when inflammatory lesions are present. There is no gold standard treatment for KP. Prevention of excessive dryness of the skin and continued moisturization are used currently as standard of care. Many topical agents such as tretinoin, ammonium lactate lotion, urea creams, tazarotene, adapalene, tacrolimus, alpha hydroxy acids and salicylic acids have been used with variable results. Sometimes topical corticosteroids are used, especially when inflammation is present. In general, KP treatments need to be continuous and complete clearance may not be possible.

Salkera emollient foam is a keratolytic foam containing 6% salicylic acid in an aqueous based emollient foam vehicle. It is different from other salicylic containing topical product in that it has been shown to produce desquamation of the stratum corneum while not effecting qualitative or quantitative changes in the structure of the viable dermis. In addition, it also contains aloe vera and anti-oxidants which help to sooth the skin. Salkera emollient foam has been used to treat several hyperkeratotic skin disorders such as KP, psoriasis, keratosis palmaris/plantaris, verrucae, icthyoses and pityriasis rubra pilaris. However, there has been no published study assessing the efficacy and safety of Salkera emollient foam in treating moderate to severe KP.

This prospective single center pilot study is designed to assess the efficacy and safety of Salkera emollient foam in treating moderate to severe KP. Patients' cosmetic acceptance of the product will also be assessed. In addition, this study is also designed to develop a validated outcome measure for assessing KP severity that can be used in future KP clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to give informed consent.
* Subject is willing and able to participate in the study as an outpatient and is willing to comply with the study requirements.
* Subject is 18 years of age or older.
* Subject has KP on 2 out of the 4 extremities.
* For each assessed extremity, subject has at least a moderate severity (≥ 3) on the Investigator Site Assessment of KP Severity.
* For each assessed extremity, subject has an aggregate score of at least 6 on the Investigator Assessment of Erythema, Roughness and Scaling.
* If subject is a female of childbearing potential, subject will have a negative urine pregnancy test at screening (week 0).
* If female, subject will be either post-menopausal for > 2 year, surgically sterile (hysterectomy or bilateral tubal ligation), or practicing one form of birth control (abstinence, oral contraceptive, estrogen patch, implant contraception, injectable contraception, IUD, diaphragm, condom, sponge, spermicides, or vasectomy of partner). Female subjects should continue to practice birth control for 1 month after the completion of study.

Exclusion Criteria:

* Subject has evidence of a clinically significant, unstable or poorly controlled medical condition as determined by the investigators/sub-investigators.
* Subject has active skin infection, atopic dermatitis or any other skin disease that will interfere with the clinical assessment of KP.
* Subject has known allergies to any ingredient of study medication.
* Subject who has used any of the following topical therapies for KP lesions within the last two weeks: topical corticosteroid, tretinoin, tazarotene, adapalene, salicylic acid, alpha-hydroxy acid, urea and/or ammonium lactate lotion.
* Subject who has been treated with UVB therapy in the last two weeks.
* Subject who has received systemic antibiotics, steroid, tacrolimus, tretinoin, isotretinoin and/or PUVA within the last 4 weeks.
* Female subjects who are pregnant (positive urine pregnancy test), breast-feeding or are considering become pregnant during the study period.
* Subject who is currently participating in another clinical trial or has completed a clinical trial within the last 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Wright State University School of Medicine, Department of Dermatology, Dayton, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening and recruitment occurred in June and July of 2009 in university dermatology clinic.
Groups:
- Treatment: Salkera foam twice a day
Period: Overall Study
Arm/Group | Treatment
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Differences Between Week 0 and Week 12 Aggregate Site Severity Score and Investigator Assessment for Site Disease Severity for All Studied Patients.
Time Frame: 12 weeks
Population: This outcome was not assessed.
Groups:
- Treatment of Study Medication: Only one study subject was enrolled. No meaning statistical analysis could be performed.
Arm/Group | Treatment of Study Medication
Number analyzed (Participants) | 0

2. Secondary Outcome: Change of Subject Assessment of Overall Disease Severity Between Week 0 and Week 12.
Description: Subject disease severity score: None (0), mild (1), mild/moderate (2), moderate (3), moderate/severe (4), severe (5).
Time Frame: 12 wks
Population: This outcome was not assessed.
Groups:
- Treatment: Only one study subject was enrolled. No meaning statistical analysis could be performed.
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No